CLINICAL TRIAL: NCT05042245
Title: The Efficacy and Safety of Ornithine Aspartic Acid Granules in Non-Alcoholic Fatty Liver Disease Against Silymarin Capsules: a Randomized, Double-Blind, Multicenter Clinical Trial
Brief Title: The Efficacy and Safety of Ornithine Aspartic Acid Granules in NAFLD Against Silymarin Capsules
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Xinhua Hospital, Shanghai Jiao Tong University School of Medicine (Other)
Collaborators: First Affiliated Hospital, Sun Yat-Sen University (Other); Beijing Ditan Hospital (Other); Beijing YouAn Hospital (Other); Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other)
Responsible Party: Principal Investigator, Jiangao Fan, Professor, Xinhua Hospital, Shanghai Jiao Tong University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: XH-19-005
Record Dates: First submitted 2021-08-24; First posted 2021-09-13 (Actual); Last update posted 2021-09-21 (Actual); Status verified 2021-09

CONDITIONS: Non-alcoholic Fatty Liver Disease
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease | interventions — Silymarin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ornithine aspartate granule group (Experimental): Patients in this group will be given aspartate ornithine granules (3 g po tid, after three meals) and silymarin capsule simulant (140 mg po bid, before breakfast and dinner).
  Interventions: Drug: Ornithine aspartate granule; Drug: Silymarin capsule simulant
- silymarin capsule group (Active Comparator): Patients in this group will be given silymarin capsule (140 mg po bid, before breakfast and dinner) and aspartate ornithine granules simulant (3 g po tid, after three meals) .
  Interventions: Drug: Silymarin capsule; Drug: Ornithine aspartate granule simulant

INTERVENTIONS:
Drug: Ornithine aspartate granule — Ornithine aspartate granules in the experimental arm.
  Arms: ornithine aspartate granule group
Drug: Silymarin capsule — Silymarin capsules in the active comparator arm.
  Arms: silymarin capsule group
Drug: Silymarin capsule simulant — Silymarin capsule simulant in the experimental arm.
  Arms: ornithine aspartate granule group
Drug: Ornithine aspartate granule simulant — Ornithine aspartate granule simulant in the active comparator arm.
  Arms: silymarin capsule group

SUMMARY:
This is a multicenter, randomized, double-blind, double-dummy, and positive control clinic trial which explores the efficacy and safety of ornithine aspartate granules in the treatment of non-alcoholic fatty liver disease against silymarin capsules. The hypothesis is that the ornithine aspartate granules have similar or better efficacy than the silymarin capsules.

ELIGIBILITY:
Inclusion Criteria:

* 1. Consistent with NAFLD diagnosis criteria, and during previous one month, the B-mode ultrasonography showed diffuse fatty liver and Fibroscan test showed that CAP value > 248 db/m;
* 2. During previous one month, serum ALT level was higher than 1.5 times the upper limit of normal.
* 3. BMI is not more than 30 kg/m2.
* 4. Voluntary to participate in the research and signed a written informed consent to comply with the trial protocol.

Exclusion Criteria:

* 1. Hereditary metabolic or autoimmune liver disease, hepatotropic and non-hepatotropic virus infection, drug/toxic/alcoholic/biliary liver injury, or any end-stage liver disease; fatty liver disease caused by one of the following reasons: total parenteral nutrition, inflammatory bowel disease, hypothyroidism, Cushing's syndrome, beta-lipoprotein deficiency and some insulin resistance (IR) related syndromes (lipid atrophic diabetes, Mauriac syndrome);
* 2. Hepatic or extrahepatic malignant tumors;
* 3. Severe heart failure or renal failure (serum creatinine > 3mg/100mL);
* 4. Allergic constitution, or allergic to amino acid drugs or to ornithine aspartate and its constituents or to silymarin;
* 5. ALT or γ-glutamyl transpeptidase (γ-GT) are greater than 5 times the upper limit of normal, or total bilirubin (TBIL) > 51 umol/L.;
* 6. Confirmed liver cirrhosis or Fibroscan test showed E value > 12.5 kilopascal (KPa);
* 7. Triglyceride > 5.6mmol/L;
* 8. Diabetes diagnosed for more than 5 years, combined with current insulin therapy or taking hypoglycemic drugs with poorly controlled condition (HbA1c > 9%).
* 9. Women who are pregnant, nursing or preparing for pregnancy;
* 10. Suspected or confirmed excessive drinking (equivalent alcohol amount: male, > 40g/d; female, > 20g/d), or history of drug abuse;
* 11. Combined use of drugs with liver protection and anti-inflammatory effects, as well as any Chinese patent medicine, Chinese herbal medicine, or health products that may have liver protection or liver damage effects;
* 12. Taking weight-loss drugs or receiving weight-loss treatment;
* 13. Situations of inappropriate participation judged by researchers.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2019-04-26 (Actual); Primary Completion 2022-06 (Estimated); Study Completion 2022-06 (Estimated)

PRIMARY OUTCOMES:
The proportion of patients whose controlled attenuation parameter (CAP) value returned to normal or changed by more than 10% | Assessed at 24 weeks

SECONDARY OUTCOMES:
The changed degree of quality-of-life measured by the Chronic Liver Disease Questionnaire (CLDQ)-NAFLD/NASH | Assessed at 4 weeks, 12 weeks, and 24 weeks
The proportion of patients whose alanine aminotransferase (ALT) level returned to normal or changed by more than 50% | Assessed at 4 weeks, 12 weeks, and 24 weeks

OTHER OUTCOMES:
The changed amount of blood ammonia | Assessed at 4 weeks, 12 weeks, and 24 weeks
  An exploratory indicator
The changed amount of body fat | Assessed at 4 weeks, 12 weeks, and 24 weeks
  An exploratory indicator of body composition analysis
The changed amount of body fat proportion | Assessed at 4 weeks, 12 weeks, and 24 weeks
  An exploratory indicator of body composition analysis
The changed amount of muscle mass | Assessed at 4 weeks, 12 weeks, and 24 weeks
  An exploratory indicator of body composition analysis

CONTACTS AND LOCATIONS:
Overall Officials: Jian G Fan, PHD, Principal Investigator — Xinhua Hospital, Shanghai Jiao Tong University School of Medicine
Locations (1):
- Xinhua Hospital, Shanghai Jiao Tong University School of Medicine, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No